CLINICAL TRIAL: NCT02845011
Title: Real-time Compression Feedback for Patients With In-hospital Cardiac Arrest: A Multi-Center Randomized Controlled Clinical Trial
Brief Title: Compression Feedback for Patients With In-hospital Cardiac Arrest
Acronym: CFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Shahid Beheshti University (Other); Tehran University of Medical Sciences (Other); East Carolina University (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, PhD, RN, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMSU CFA Prospective
Record Dates: First submitted 2016-07-21; First posted 2016-07-26 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Cardiopulmonary Arrest; Cardiopulmonary Resuscitation
Keywords: Cardio first angle; CPR; Cardiopulmonary Arrest; Clinical trial
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The clinical provider was not involved in the study. S(he) was not blind during the resuscitation as they could see device, and it was not considered ethical to employ a sham device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Audiovisual compression feedback (Experimental): Cardiopulmonary resuscitation according to international guidelines with chest compressions performed with real-time audiovisual feedback using the Cardio First Angel™ (CFA; INOTECH, Nubberg, Germany) device.
  Interventions: Device: Audiovisual compression feedback
- Standard chest compression (Active Comparator): Cardiopulmonary resuscitation according to international guidelines with standard manual chest compression
  Interventions: Other: Standard Manual Chest Compression

INTERVENTIONS:
Device: Audiovisual compression feedback — The Cardio First Angel™ (CFA; INOTECH, Nubberg, Germany) is a handheld device consisting of three components. The rescuer-side has a red palm-sized push-button with a pictogram illustrating proper use. The center unit is composed of a stable plastic base containing an arrangement of springs, and the patient-side consists of liquid-absorbent polyurethane foam. Application of 400 ± 30 Newtons of force results in an audible click alerting the rescuer to cease compression, and an additional click on decompression alerts the rescuer to resume compression.
  Other Names: Cardio First Angel™
  Arms: Audiovisual compression feedback
Other: Standard Manual Chest Compression — Cardiopulmonary resuscitation according to published international guidelines.
  Arms: Standard chest compression

SUMMARY:
A prospective, randomized, controlled, parallel study was conducted in patients undergoing resuscitation with chest compression for in-hospital cardiac arrest (IHCA) in the mixed medical-surgical ICU's of 8 academic tertiary care hospitals in Iran. Patients randomized into 2 groups: 1) standard chest compression, 2) chest compression with real-time audio-visual feedback using the Cardio First Angel™ (CFA; INOTECH, Nubberg, Germany) device. The primary outcome was sustained return of spontaneous circulation (ROSC). Secondary outcomes were survival to ICU and hospital discharge, incidence of sternum and rib fractures.

DETAILED DESCRIPTION:
A prospective, randomized, controlled, parallel study was conducted in patients undergoing resuscitation with chest compression for in-hospital cardiac arrest (IHCA) in the mixed medical-surgical ICU's of 8 academic tertiary care hospitals in Iran. Patients randomized into 2 groups: 1) standard chest compression, 2) chest compression with real-time audio-visual feedback using the Cardio First Angel™ (INOTECH, Nubberg, Germany) device. Randomization accomplished using Random Allocation Software© (RAS; Informer Technologies, Inc., Madrid, Spain). Crossover was not allowed. The patient and data analyzer were blinded. The clinical provider was not blinded. The primary outcome was sustained return of spontaneous circulation (ROSC). Secondary outcomes were survival to ICU and hospital discharge, incidence of sternum and rib fractures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to the intensive care unit (ICU)
* Full-code status
* Informed consent was obtained from the patient, legal guardian, or healthcare surrogate upon ICU admission (prior to cardiac arrest event)

Exclusion Criteria:

* Patients with any limitation of code status including but not limited to "no code" or"do not resuscitate" (DNR) and"do not intubate" (DNI), were excluded from study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Sustained Return of Spontaneous Circulation | 30 minutes after completion of cardiopulmonary resuscitation
  Return of spontaneous circulation

SECONDARY OUTCOMES:
Survival to ICU discharge | through ICU discharge, usually 15-35 days
  Survival to first or only ICU discharge
Survival to Hospital Discharge | through study completion, usually 30-45 days
  Survival to Hospital Discharge
Fractures | through study completion, usually less than 60 days
  Number of rib or sternum fractures

CONTACTS AND LOCATIONS:
Overall Officials: Amir Vahedian-azimi, PhD, RN, Principal Investigator — Baqiyatallah Universiy of Medical Sciences

REFERENCES:
- [Derived] Goharani R, Vahedian-Azimi A, Farzanegan B, Bashar FR, Hajiesmaeili M, Shojaei S, Madani SJ, Gohari-Moghaddam K, Hatamian S, Mosavinasab SMM, Khoshfetrat M, Khabiri Khatir MA, Miller AC; MORZAK Collaborative. Real-time compression feedback for patients with in-hospital cardiac arrest: a multi-center randomized controlled clinical trial. J Intensive Care. 2019 Jan 22;7:5. doi: 10.1186/s40560-019-0357-5. eCollection 2019. PMID 30693086